CLINICAL TRIAL: NCT02512783
Title: Decreasing Propofol Injection Pain by Pre-Treatment With Lidocaine in Pediatric Procedural Sedation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis indicated treatment was effective and statistically significant
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1302-019
Record Dates: First submitted 2013-08-15; First posted 2015-07-31 (Estimated); Results first posted 2016-06-17 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-06

CONDITIONS: Pain
Keywords: Propofol; Lidocaine; Intravenous propofol
MeSH Terms: conditions — Pain | interventions — Lidocaine; Saline Solution; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Active Comparator): Administration of 1ml of pre-treatment 1% lidocaine immediately prior to propofol induction.
  Interventions: Drug: Lidocaine; Drug: Propofol
- Normal Saline (Placebo Comparator): Administration of 1ml of pre-treatment normal saline immediately prior to propofol induction.
  Interventions: Drug: Normal Saline; Drug: Propofol

INTERVENTIONS:
Drug: Lidocaine — Administration of 1ml of pre-treatment 1% lidocaine 1-minute prior to sedation
  Other Names: Xylocaine
  Arms: Lidocaine
Drug: Normal Saline — Administration of 1ml of pre-treatment normal saline 1-minute prior to sedation
  Arms: Normal Saline
Drug: Propofol — Intravenous administration of propofol according to standard care to sedate patient.
  Other Names: Diprivan; Fresenius Propoven

SUMMARY:
This is a double blind, randomized, controlled study. The sedationist performing the sedation procedure will inject the appropriate amount of either a 1% Lidocaine solution or a placebo before the administration of Propofol. A research staff will observe the patient simultaneously with the induction of Propofol to determine the patient's pain level, as measured by the Face, Legs, Activity, Cry, Consolability (FLACC) scale. The purpose of this study is to determine the efficacy of premedication with 1% Lidocaine in decreasing the burning sensation caused by intravenous Propofol.

DETAILED DESCRIPTION:
Propofol is a short-acting, intravenously administered anesthetic. It has become a popular choice for procedural sedation in both children and adults. Despite its many advantages, Propofol is associated with a burning sensation during injection. Propofol pain begins within the first few seconds after administration and often lasts approximately 10-20 seconds until the patient is asleep. Lidocaine is often used in an attempt to reduce Propofol injection pain, but neither its delivery mode nor concentration has been standardized.

The purpose of this study is to determine the efficacy of premedication with 1% Lidocaine in decreasing the burning sensation caused by intravenous Propofol.

This is a double blind, randomized, controlled study. The sedationist performing the sedation procedure will inject the appropriate amount of either a 1% Lidocaine solution or a placebo before the administration of Propofol. A research staff will observe the patient simultaneously with the induction of Propofol to determine the patient's pain level, as measured by the FLACC scale.

ELIGIBILITY:
Inclusion Criteria:

* age 2 months to 17 years
* patient already scheduled for procedural sedation with propofol
* sedation procedure to be performed by a sedationist from Children's Respiratory and Critical Care Specialists

Exclusion Criteria:

* patients who are not receiving deep sedation with propofol
* patients with allergy or other contraindication to lidocaine administration
* patients with central venous catheters as propofol does not burn when given centrally
* patients being premedicated with an analgesic other than nitrous oxide or 1% lidocaine
* patients weighing less than 5 kg to prevent any risk of inadvertent lidocaine overdose.

Ages: 2 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 171 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Didima Mon-Sprehe, MD, Principal Investigator — Children's Hospitals and Clinics of Minnesota
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lidocaine | Normal Saline
Started | 96 | 75
Completed | 96 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine | Normal Saline | Total
Number analyzed (Participants) | 96 | 75 | 171
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 96 | 75 | 171
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 35 | 75
  Male | 56 | 40 | 96

OUTCOME MEASURES:

1. Primary Outcome: Change in FLACC (Face, Legs, Activity, Cry, Consolability) Score
Description: The FLACC scale measures pain in children aged 2m-7y. The scale ranges from 0-10 with 0 being no pain. The total score out of 10 is based on 5 pieces of criteria, and each criteria is scored as either 0, 1, or 2. Scores on individual criteria are summed up to give a total score. Higher values represent a worse outcome of more pain. FLACC scores will be compared pre- and post-propofol induction to assess the change in FLACC score for each arm.
Time Frame: 1 minute before propofol induction compared to 1 minute following propofol induction
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Normal Saline
Number analyzed (Participants) | 96 | 75
units on a scale | .82 (2.357) | 2.43 (3.268)

2. Secondary Outcome: Parental Assessment of Child's Pain on a Visual Analog Scale
Time Frame: Immediately following propofol injection
Population: This data was not collected.
Arm/Group | Lidocaine | Normal Saline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Lidocaine | Normal Saline
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/75
Other Adverse Events (participants affected / at risk) | 0/96 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes